CLINICAL TRIAL: NCT05849298
Title: An International Prospective Open-label, Multi-center, Randomized, Non-comparative Phase II Study of Lutetium [177Lu] Vipivotide Tetraxetan (AAA617) Alone and Lutetium [177Lu] Vipivotide Tetraxetan (AAA617) in Combination With Androgen Receptor Pathway Inhibitors in Patients With PSMA PET Scan Positive Castration-Resistant Prostate Cancer
Brief Title: A Phase II Study of AAA617 Alone and AAA617 in Combination With ARPI in Patients With PSMA PET Scan Positive CRPC
Acronym: PSMACare
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617B12203; 2022-503040-41-00 (Other: EU CT Number)
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasm
Keywords: Prostate-specific membrane antigen (PSMA); Lutetium [177Lu] vipivotide tetraxetan (AAA617); Androgen Receptor Pathway Inhibitors (ARPI); Enzalutamide; Darolutamide; Apalutamide; Castration Resistant Prostate Cancer; Androgen Deprivation Therapy; gallium [68Ga] gozetotide (AAA517); piflufolastat F 18
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium; Lutetium-177; Pluvicto; gallium 68 PSMA-11; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Intervention Model Description: No cross-over allowed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive 7.4 GBq (+/- 10%) of AAA617 (Lutetium [177Lu] vipivotide tetraxetan) once every 6 weeks for 6 cycles. ADT must be ongoing; Best supportive care is allowed.
  Interventions: Drug: AAA617; Drug: AAA517; Drug: Piflufolastat F 18; Drug: ADT; Other: Best supportive care
- Arm B (Experimental): Participants will receive 7.4 GBq (+/- 10%) of AAA617 (Lutetium [177Lu] vipivotide tetraxetan) once every 6 weeks for 6 cycles. In addition of SOC (ADT plus choice of ARPI as per physician's decision), Best supportive care is allowed.
  Interventions: Drug: AAA617; Drug: AAA517; Drug: Piflufolastat F 18; Drug: ARPI; Drug: ADT; Other: Best supportive care

INTERVENTIONS:
Drug: AAA617 — Administration intravenously once every 6 weeks (1 cycle) for 6 cycles
  Other Names: Lutetium [177Lu] vipivotide tetraxetan; 177Lu-PSMA-617
Drug: AAA517 — Single intravenous dose of approx. 150 Megabecquerel (MBq) prior PSMA-PET scans
  Other Names: 68Ga-PSMA-11
Drug: Piflufolastat F 18 — Single intravenous dose of approx. 333 Megabecquerel (MBq) prior PSMA-PET scans
Drug: ARPI — Enzalutamide, Darolutamide, Apalutamide as prescribed by the local investigator
  Arms: Arm B
Drug: ADT — as prescribed by the local investigator
Other: Best supportive care — as prescribed by the local investigator

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AAA617 alone (Lutetium [177Lu] vipivotide tetraxetan) and in combination with an Androgen Receptor Pathway Inhibitors (ARPI) in participants with PSMA-positive, castration-resistant prostate cancer and no evidence of metastasis in conventional imaging (CI) (i.e., CT/MRI and bone scans). Approximately 80 participants will be randomized.

ELIGIBILITY:
Key Inclusion criteria

* Participants must be adults ≥ 18 years of age with signed informed consent prior to participation to study
* Histologically or cytologically confirmed prostate cancer
* Participants must have ongoing androgen deprivation therapy with a GnRH agonist/antagonist or prior bilateral orchiectomy at the time of randomization. Intermittent administration of ADT is accepted before randomization if criterion for serum testosterone is met
* Castrate level of serum testosterone (< 1.7 nmol/l [50 ng/dl]) on GnRH agonist or antagonist therapy (continuous/intermittent) or after bilateral orchiectomy prior to randomization
* Participants must have evidence of PSMA-positive disease (N1 or M1) as seen on a AAA517 or piflufolastat F 18 PET/CT scan at baseline as determined by Blinded Independent Central Review (BICR) based on the methodology proposed in the Prostate Cancer Molecular Imaging Standardized Evaluation (PROMISE) (Eiber et al 2018). Participants with M1 disease only on PSMA PET scan are allowed to participate
* Participants must have a negative conventional imaging for M1 disease.
* Participants must have adequate organ functions: bone marrow reserve, hepatic & renal

Key Exclusion criteria

* Prior or present evidence of metastatic disease as assessed by CT/MRI locally for soft tissue disease and whole-body radionuclide bone scan for bone disease. Exception: Participants with pelvic disease may be eligible (e.g., participants with enlarged lymph nodes below the bifurcation of common iliac arteries (N1))
* Unmanageable concurrent bladder outflow obstruction or urinary incontinence. Note: participants with bladder outflow obstruction or urinary incontinence, which is manageable with best available standard of care (incl. pads, drainage) are allowed
* Active clinically significant cardiac disease; history of seizure or condition that may pre-dispose to seizure which may require treatment with surgery or radiation therapy
* Prior therapy with: second generation anti-androgens (e.g., enzalutamide, apalutamide and darolutamide) < 3 months before randomization; CYP17 inhibitors (e.g., abiraterone acetate, orteronel, galeterone) < 3 months before randomization; ketoconazole (short duration ketoconazole treatment (<28 days) is permitted); radiopharmaceutical agents (e.g., Strontium-89) if wash-out period of at least 3 months is not completed, PSMA-targeted radioligand therapy; immunotherapy (e.g., sipuleucel-T); chemotherapy, except if administered in the adjuvant/neoadjuvant setting, completed > 2 years before randomization; any other investigational agents for CRPC; use of estrogens, 5-α reductase inhibitors (finasteride, dutasteride), other steroidogenesis inhibitors (aminoglutethimide) or first-generation anti-androgens (bicalutamide, flutamide, nilutamide, cyproterone) within 28 days before randomization; radiation therapy (external beam radiation therapy [EBRT] and brachytherapy within 28 days before randomization
* Other concurrent cytotoxicity chemotherapy, immunotherapy, radioligand therapy, poly adenosine diphosphate-ribose polymerase (PARP) inhibitor, biological therapy or investigational therapy

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer study
Enrollment: 47 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2028-04-07 (Estimated); Study Completion 2030-05-18 (Estimated)

PRIMARY OUTCOMES:
PSA response | From randomization until PSA nadir value of =< 0.2 ng/mL that is confirmed by a second (the next) PSA measurement >= 4 weeks later, up to 5 years
  PSA response is defined as the time of PSA nadir value of =< 0.2 ng/mL is confirmed by a second (the next) PSA measurement at least 4 weeks later

SECONDARY OUTCOMES:
Metastatic Free Survival (MFS) | From date of randomization until date of progression or date of death whichever occurs first, up to 5 years
  MFS is defined as the time from date of randomization to the first evidence of radiographically detectable bone or soft tissue distant metastasis by conventional imaging using RECIST 1.1 or death.
Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, up to 5 years
  rPFS is defined as the time from the date of randomization to the date of first documented radiographic disease progression by conventional imaging assessed using RECIST 1.1 or death.
Overall Survival (OS) | From date of randomization until date of death from any cause, up to 5 years
  OS defined as date of death due to any cause
second Progression Free Survival (PFS2) | From date of randomization until date of second progression or date of death from any cause, whichever comes first, assessed up to 5 years
  PFS2 defined as time from the date of randomization to the date of first documented disease progression by investigator's assessment (PSA, radiographic, symptomatic, or any combination) on next line of therapy subsequent to MFS event or death due to any cause, whichever occurs first
Time to symptomatic progression | From date of randomization until development of a symptomatic skeletal event, new systemic anti-cancer therapy, surgical intervention or radiation therapy, whichever occurs first, up to 5 years
  Time to symptomatic progression will be defined as the time from the date of randomization to the date of first documented event for any of the following:
  * Development of a symptomatic skeletal event (SSE)
  * Pain progression or worsening of disease-related symptoms requiring initiation of a new systemic anti-cancer therapy
  * Development of clinically significant symptoms due to loco-regional tumor progression requiring surgical intervention or radiation therapy
Time to initiation of cytotoxic chemotherapy | From the date of randomization to the date of first documented dose of new cytotoxic chemotherapy administered to the participant, up to 5 years
  Time to initiation of cytotoxic chemotherapy will be defined as the time from the date of randomization to the date of first documented dose of new cytotoxic chemotherapy being administered to the participant
Time to first symptomatic skeletal event (TTSSE) | From the date of randomization to the date of the first new symptomatic pathological bone fracture, spinal cord compression, orthopedic surgical intervention, radiation therapy or death due to any cause, whichever occurs first, up to 5 years
  TTSSE is defined as the time from the date of randomization to the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death due to any cause, whichever occurs first
Time to distant metastasis development | From the date of randomization to the date of first evidence of radiographically detectable bone or soft tissue distant metastasis, up to 5 years
  Time to distant metastasis development is defined as the time from the date of randomization to the date of first evidence of radiographically detectable bone or soft tissue distant metastasis by conventional imaging using RECIST 1.1
Time to local radiological progression | From the date of randomization to the date of first documented local radiographic disease progression, up to 5 years
  Time to local radiological progression is defined as the time from the date of randomization to the date of first documented local radiographic disease progression by conventional imaging using RECIST 1.1
Time to initiation or change in therapy | From the date of randomization to the date of first dose of a new / change in therapy, up to 5 years
  Time to initiation or change in therapy is defined as the time from the date of randomization to the date of first documented dose of a new / change in therapy being administered to the participant
Time to PSA response | From randomization to PSA response, up to 5 years
  Time to PSA response is calculated as the time from randomization to PSA response with a PSA nadir value of =< 0.2ng/mL.
PSA50 response | From date of randomization until end of efficacy follow-up, up to 5 years
  PSA50 response is defined as the proportion of participants who have a >= 50% decrease in PSA from baseline that is confirmed by a second (the next) PSA measurement >= 4 weeks later
PSA90 response | From date of randomization until end of efficacy follow-up, up to 5 years
  PSA90 response is defined as the proportion of participants who have a >= 90% decrease in PSA from baseline that is confirmed by a second (the next) PSA measurement >= 4 weeks later
Functional Assessment of Cancer Therapy - Prostate (FACT-P) | From date of randomization until end of efficacy follow-up, up to 5 years
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Functional Assessment of Cancer Therapy - Radiotherapies (FACT-RNT) Questionnaire | From date of randomization until end of efficacy follow-up, up to 5 years
  The FACT-RNT is assessing treatment-related symptoms of special interest/associated with Radionuclides Therapies. The FACT-RNT contains 15 items assessing dry mouth, dry eyes, difficulty urinating, nausea, vomiting, diarrhea, constipation, loss of appetite, fatigue, impact of fatigue, pain, bone pain, pain interference, bothered by of side effects of treatment and isolation due to illness or treatment.
Brief Pain Inventory - Short Form (BPI-SF) Questionnaire | From date of randomization until end of efficacy follow-up, up to 5 years
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (16):
  - Urology Associates of Mobile, Mobile, Alabama
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University Of Florida, Jacksonville, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Urology Of Indiana, Indianapolis, Indiana
  - Unity Point Clinic, Des Moines, Iowa
  - Urology Cancer Center PC, Omaha, Nebraska
  - Associated Med Professionals of NY, Syracuse, New York
  - Oregon Urology Institute, Springfield, Oregon
  - Wellspan York Hospital, York, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinic of North Texas, Dallas, Texas
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - Rio Grande Urology, El Paso, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Health San Antonio Mays Cancer Center, San Antonio, Texas
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Canada (3):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Olomouc, Czechia
- France (5):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (3):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Rostock
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Arnhem, Gelderland, Netherlands
- Poland (2):
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (6):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.